CLINICAL TRIAL: NCT05307484
Title: Effects of a Serious Game on Knowledge, Attitude and Practice in Vector Control and Dengue Prevention Among Adults in Primary Care: A Randomized Controlled Trial
Brief Title: Effects of a Serious Game on Knowledge, Attitude and Practice in Vector Control and Dengue Prevention Among Adults in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SingHealth Polyclinics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020/3091
Record Dates: First submitted 2022-03-18; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Dengue
Keywords: Serious game; Dengue prevention; Primary care
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial was conducted among volunteer adults who were visiting a regional primary care clinic in Sengkang, Singapore. 400 participants were randomly allocated to receive information regarding dengue prevention from either playing a serious game (intervention) or visiting a dengue prevention website (control). Before and after receiving information on dengue prevention, participants completed a self-administered questionnaire within a 2-week interval to assess the knowledge, attitude and practice (KAP) score and their interest to vaccinate against dengue. Participants, who played serious game, evaluated the game with the Systems Usability Score (SUS).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomization sequence was prepared by the bio-statistician who was not involved in the enrollment of the participants. The outcome data was collected via a participant-administered questionnaire on an online secured platform, without contact with the study members. All data were de-identified and the statistical analysis was performed by the bio-statistician, who was blinded to group allocation, only after the completion of enrollment of all participants. The principal investigator was not involved in the enrollment or randomization process of participants in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serious game group (Experimental): Participants in the intervention group installed a mobile application, 'Sam's Mozzie Adventure'. This is a locally designed serious game which was co-created between SingHealth Polyclinics and AI Innovation Labs (AI2 Labs) Private Limited, specifically for this study. The principal investigator reviewed existing publicly available information on dengue prevention, including those on the National Environmental Agency (NEA) 'Stop Dengue' website, and provided the relevant content and pedagogical knowledge to the team of app developers from AI2 Labs. After creating the syllabus, the developers deployed their technological knowledge to integrate the dengue prevention information into the serious game. The participants were instructed to complete playing this serious game within 2 weeks.
  Interventions: Other: Serious game
- Dengue prevention website group (Active Comparator): The control group accessed the NEA 'Stop Dengue' website which contained dengue prevention information in the forms of online articles, posters and video. The participants were instructed to complete reading the online resources within 2 weeks.
  Interventions: Other: Dengue prevention website

INTERVENTIONS:
Other: Serious game — This is a serious game in the form of a mobile application, designed to educate adults on dengue prevention.
  Other Names: Sam's Mozzie Adventure
  Arms: Serious game group
Other: Dengue prevention website — This is a website containing information regarding dengue prevention.
  Other Names: National Environmental Agency 'Stop Dengue' website
  Arms: Dengue prevention website group

SUMMARY:
Dengue can be mitigated by both vector control and vaccination. Serious games in healthcare can be used to raise the community awareness of vector control in dengue prevention in a simulated interactive learning environment, by motivating serious game participants to optimise their own performance and influence their behaviour. The results show a specially designed serious game can better engage local residents by raising their awareness in vector control and proactiveness in dengue prevention. At least 8 out of 10 participants were willing to be vaccinated against dengue if they knew of the availability of a safe and effective vaccine.

DETAILED DESCRIPTION:
Study design: From March to August 2021, a single-centre randomised controlled trial was conducted to determine the effectiveness of playing a serious game (intervention) in improving the KAP of participants in vector control and dengue prevention compared to those who viewed a dengue prevention website (control).

Study site: This study was conducted at a regional public primary care clinic (Polyclinic) in Sengkang. Sengkang Polyclinic is located in Sengkang Community Hub, which is an amenity centre in Sengkang, within the North-East region of Singapore. Sengkang is also a residential town, which is the second most populous in the region, being home to 244,600 residents in 2019.

Sample size calculation: To determine the effect of serious game in the literacy level of adults in preventing dengue in Singapore, the sample size was computed based on the study by Nurul Akmar Ghani et al, in which the significant difference in mean and standard deviation of knowledge scores were 14.55 (3.09) and 15.41 (2.75) respectively between the compared groups. To obtain a sample size with 95% confidence level and 80% power for this study, a minimum of 182 participants per group was required. With a possible drop out of 10%, the sample size was increased to 200 per group.

Recruitment and consent process: Recruitment posters, containing registration details of the study, were placed within the clinic's premises from March to August 2021. Adults who were interested to join the study voluntarily could approach the clinical research coordinators (CRCs), who would screen them for eligibility, explained the study intent and procedure to them in a designated room within the study site. The CRCs were trained by the principal investigator to provide adequate information and address relevant concerns or queries from the participants prior to the start of this study. The latter were informed about the purpose and content of the study based on the approved participant information sheet. After clarifying their doubts and queries, every eligible participant endorsed their written informed consent before randomization.

Randomization: The randomization sequence was created by the biostatistician using computer generated random numbers in a 1:1 ratio. Random permuted blocks were used to ensure equal number in each group. The randomization sequence was concealed in sequentially numbered, opaque, sealed envelopes by the principal investigator (PI) at the study site, and stored in a secured location that was accessible only by the research assistants. Blinding was not possible for the participants and the CRCs, as the intervention group would be required to download an application into the mobile phone. Both the biostatistician and PI were not involved in the enrolment or randomization process of participants in this study.

Study procedure: The KAP assessment instrument was adapted from a previous study conducted by Nurul Akmar Ghani et al.

Participants in both groups completed the first (baseline) questionnaire via a secured online platform, Form.sg. Form.sg was used to create online questionnaires that capture classified data for this study. The platform does not store participants' response data in its servers and all responses are sent directly to the study team's dedicated email address.

Participants in the intervention group installed a mobile application, 'Sam's Mozzie Adventure' and were instructed to complete the game within 2 weeks.

Participants in the control group accessed the National Environmental Agency 'Stop Dengue' website and were instructed to complete reading the dengue prevention information within 2 weeks.

Both groups completed the second questionnaire, containing the KAP assessment and a question pertaining to individual's interest to vaccinate against dengue, within 2 weeks after the intervention. In addition, participants in the serious game group evaluated the game with the adapted Systems Usability Score.

Analysis: The knowledge, attitude and practice scores varied from 0-16, 0-15, 0-15 respectively, with a maximum score of 46 points. The highest achievement attained by the participants in serious game group were measured by the number of stars awarded in-game, which varied from 0-48 stars. The data were audited and errors were rectified before analyses. Descriptive statistics in terms of frequency (n), percentage (%), mean and standard deviations (SD) were used to express the data. The socio-demographic variables between the two groups were compared using Chi-Square test for categorical variables and independent t-test for continuous variables. Independent t-test was used to compare the baseline, follow up and change in KAP scores between the control and intervention group. Paired t-test was used to determine the difference in scores from baseline and follow up. The Spearman's correlation was used to determine the association between change scores and maximum game stars awarded in the intervention group. SUS score was presented in frequency and percentages. A p-value of less than 0.05 is considered statistically significant. All analyses were performed using IBM SPSS 27.0.

ELIGIBILITY:
Inclusion Criteria:

* Adult who is visiting Sengkang Polyclinic.
* Able to understand English.
* Has a mobile phone which was compatible with the serious game and willing to download and attempt the serious game.
* Able to complete questionnaires on the online secured platform, Form.sg.

Exclusion Criteria:

* Adult who is not able to use a mobile phone due to physical or cognitive impairments.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Change of knowledge, attitude and practice (KAP) assessment score on dengue fever prevention | Change from baseline KAP score at 2 weeks (or within 2 weeks after completion of intervention)
  This outcome is measured via a participant-administered questionnaire which was used and validated in previous regional studies. It is divided into 3 sections: (1) knowledge (16 items), (2) attitude (15 items), (3) practice (15 items) in preventing dengue.
  The minimum and maximum values of this questionnaire are 0 and 46 respectively. A higher score indicates a better outcome.

SECONDARY OUTCOMES:
Change of interest to vaccinate against Dengue | Change from baseline Dengue vaccination interest at 2 weeks (or within 2 weeks after completion of intervention)
  This outcome is measured via a participant-administered questionnaire. It consists of 1 section: (1) interest to vaccinate against Dengue (1 item).
  A higher proportion of participants indicating interest to vaccinate against Dengue indicates a better outcome.
System Usability Scale (SUS) score of serious game | At 2 weeks from start of study (or within 2 weeks after completion of intervention by the serious game group)
  This outcome is measured via a participant-administered questionnaire. It is modified from the validated SUS template to evaluate the usability of this serious game. The SUS has 10 statements, and a 5-point Likert scale is used to indicate the participant's agreement with the statements.
  The response of each participants is collated and a standardized formula is applied to calculate the final SUS score. A score above 68 is above average and scores below 68 is below average in terms of system usability.
  A score of less than 68 indicates that the participants may have less than average user experience with the serious game.

CONTACTS AND LOCATIONS:
Overall Officials: Alon Tan, Principal Investigator — SingHealth Polyclinics
Locations (1):
- SingHealth Polyclinics - Sengkang, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No